CLINICAL TRIAL: NCT03891875
Title: A Phase 2 Randomized, Double-Masked, Placebo-Controlled Clinical Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Elamipretide in Subjects With Age-Related Macular Degeneration With Non-central Geographic Atrophy
Brief Title: ReCLAIM-2 Study to Evaluate Safety,Efficacy & Pharmacokinetics of Elamipretide in Subjects With AMD With Non-central GA
Acronym: ReCLAIM-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIAM-202
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Age-related Macular Degeneration
Keywords: AMD; Macular degeneration; non-central geographic atrophy; MTP-131; elamipretide
MeSH Terms: conditions — Macular Degeneration | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elamipretide (Experimental): Once daily 40 mg subcutaneous injection of elamipretide using the elamipretide delivery system for 48 weeks followed by a 4 week follow-up period.
  Interventions: Combination Product: Subcutaneous elamipretide through the elamipretide delivery system
- Placebo (Placebo Comparator): Once daily subcutaneous injection of placebo using the elamipretide delivery system for 48 weeks followed by a 4 week follow-up period.
  Interventions: Combination Product: Subcutaneos placebo through the elamipretide delivery system

INTERVENTIONS:
Combination Product: Subcutaneous elamipretide through the elamipretide delivery system — Subjects will be randomized in a 2:1 ratio to receive either elamipretide or placebo through the elamipretide delivery system. Subjects will dose daily for up to 48 weeks.
  Other Names: elamipretide; MTP-131; Bendavia
  Arms: Elamipretide
Combination Product: Subcutaneos placebo through the elamipretide delivery system — Subjects will be randomized in a 2:1 ratio to receive either elamipretide or placebo through the elamipretide delivery system. Subjects will dose daily for up to 48 weeks.
  Arms: Placebo

SUMMARY:
A randomized, double-masked, placebo-controlled study to evaluate the safety, efficacy and pharmacokinetics of elamipretide in subjects with Age-Related Macular Degeneration with non-central Geographic Atrophy.

DETAILED DESCRIPTION:
This was a randomized, double-masked, placebo controlled study using three periods to evaluate the safety, efficacy and pharmacokinetics of elamipretide in subjects with Age-Related Macular Degeneration with non-central Geographic Atrophy. The total duration of subject participation was up to 54 weeks, including a Screening Period (≤2 weeks), Treatment Period (48 weeks), and Follow-up (4 weeks). 176 eligible subjects were randomized in a 2:1 ratio (elamipretide:placebo) to receive 40 mg elamipretide or placebo. The study drug (i.e., elamipretide or placebo) was administered once daily via SC injection using the elamipretide delivery system during the 48 week Treatment Period. After completion of the 48-week Treatment Period subjects continued to be monitored for safety during the 4-week Follow-up Period and an end of study (EOS) Follow-up Visit was conducted at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 55 years of age with at least 1 eye with AMD with non-central GA as determined by FAF.

Ocular conditions-study eye

* GA in the study eye at the Screening Visit may be multi-focal, but the cumulative GA lesion and size must:

  1. be ≥ 0.05 mm2 and ≤ 10.16 mm2 and
  2. reside completely within the FAF 30 or 35 degree image.
  3. must be at least 150 μm from foveal center with preserved outer retinal structural details
* No evidence of CNV by history, OCT or FA in the study eye.
* BCVA by Early Treatment Diabetic Retinopathy Study (ETDRS) score of ≥ 55 letters (Snellen equivalent ≥ 20/70) in the study eye at the Screening Visit and Baseline Visit.
* LL BCVA by ETDRS score of ≥ 10 letters in the study eye at the Screening Visit and Baseline Visit.
* LL VA deficit (defined as difference the between BCVA and LL BCVA) of > 5 letters in the study eye at Screening and Baseline Visits.
* The fellow eye may have any of the following: no AMD, AMD without GA, AMD with GA, CNV AMD, or central GA. Ongoing treatment with anti-angiogenic therapies in the fellow eye is allowable.
* Sufficiently clear ocular media, adequate pupillary dilation, fixation to permit quality fundus imaging, and ability to cooperate sufficiently for adequate ophthalmic visual function testing and anatomic assessment in the study eye.

Systemic and general criteria

Exclusion Criteria:

Ocular conditions-study eye

* The absence of observable hyper-FAF at the margins of the GA in the study eye(only for lesions ≥ 0.25mm2)
* Atrophic retinal disease of causality other than AMD including myopia-related maculopathy and monogenetic macular dystrophies including pattern dystrophy and adult-onset Stargardt disease in the study eye.
* Presence or diagnosis of exudative AMD or CNV in the study eye.
* Presence of retinal vein occlusion in the study eye.
* Presence of diabetic retinopathy (a history of diabetes mellitus without retinopathy is not a criterion for exclusion) in either eye.
* Presence of vitreous hemorrhage in the study eye.
* History of retinal detachment in the study eye.
* History of macular hole (stages 2 to 4) in the study eye.
* Presence of an epiretinal membrane that causes distortion of the retinal contour in the study eye.
* Presence of vitreomacular traction in the study eye.
* At the Screening Visit, advanced glaucoma resulting in a cup to disc ratio of > 0.8 in the study eye.
* History of glaucoma filtration surgery or uncontrolled glaucoma defined as IOP > 22 mmHg at baseline despite anti-glaucoma treatment with or without topical anti-hypertensive eye drops in the study eye OR currently using > 2 medications (note: combination medications count as 2 medications).
* Presence of visually significant cataract OR presence of significant posterior capsular opacity in the setting of pseudophakia. Significant cataract is defined as > +2 nuclear sclerosis based upon the scale below or any Posterior Subcapsular Cataract in the study eye. The Sponsor, or its designee, will supply the trial sites with a copy of the standard photographs.
* Presence of significant keratopathy or any other media or corneal opacity that would cause scattering of light or alter visual function, especially in LL conditions in the study eye.
* Ocular incisional or laser surgery (including cataract surgery) in the study eye within 90 days before Day 1.
* Yag laser capsulotomy in the study eye within 30 days before Day 1.
* Aphakia in the study eye.
* History of vitrectomy surgery, submacular surgery, or any vitreoretinal surgery in the study eye.
* Prior treatment with Visudyne® (verteporfin) ocular photodynamic therapy, external-beam radiation therapy (for intraocular conditions), or transpupillary thermotherapy in the study eye.
* History of subthreshold laser treatment or other forms of photobiomodulation for AMD in the study eye.
* Intravitreal drug delivery in the past 60 days or 5-half-lives of the injected drug whichever is longer (e.g., intravitreal corticosteroid injection, anti angiogenic drugs, or device implantation) in the study eye.
* Current use of medications known to be toxic to the lens, retina, or optic nerve (e.g., deferoxamine, chloroquine/hydroxychloroquine [Plaquenil®], tamoxifen, phenothiazines, ethambutol, digoxin, and aminoglycosides) from the Screening Visit through the completion of the trial.

Ocular conditions--either eye

* History of herpetic infection in either eye.
* Concurrent disease in either the study eye or fellow control eye that could require medical or surgical intervention during the study period.
* Active uveitis and/or vitritis (grade trace or above) in either eye.
* History of idiopathic or autoimmune-associated uveitis in either eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.

Systemic conditions.

* Known to be immunocompromised or receiving systemic immunosuppression for ≥ 4 consecutive weeks prior to screening.
* Any disease or medical condition that in the opinion of the Investigator would prevent the subject from successfully participating in the study or might confound study results.

General

* Participation in other investigational drug or device clinical studies within 30 days of enrollment and/or planning to participate in any other investigational drug or device clinical studies within 30 days of study completion.
* History of allergy to fluorescein that is not amenable to treatment.
* Creatinine clearance of ≤ 30 mL/min at the Screening Visit (using Modification of Diet in Renal Disease Study formula).
* Inability to comply with study or follow-up procedures.
* Inability to obtain color fundus photograph, FAF, and FA of sufficient quality to be analyzed and interpreted.
* Active malignancy or any other cancer from which the subject has been cancer-free for < 2 years.
* History of allergic reaction to the investigational drug or any of its components.
* Prior treatment with Elamipretide.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sathyanarayana, Study Director — Stealth BioTherapeutics
Locations (36):
- United States (36):
  - Associated Retina Consultants, Ltd., Peoria, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Arizona Retina & Vitreous Consultants, Phoenix, Arizona
  - Global Retina Institute, Scottsdale, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Institute of California Medical Group, Palm Desert, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - MedEye Associates, Miami, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - The Retina Care Center, Baltimore, Maryland
  - Cumberland valley retina consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Specialty Eye Institute, Jackson, Michigan
  - Retina Center of New Jersey LLC, Bloomfield, New Jersey
  - New Jersey Retina, Teaneck, New Jersey
  - Retina Associates of Western New York, Rochester, New York
  - Duke Eye center, Durham, North Carolina
  - Sterling Research Group, Cincinnati, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Retina Northwest, P.C, Portland, Oregon
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Tennessee Retina, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Retina Consultants of Houston, Katy, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - University of Virginia, Department of Ophthalmology, Charlottesville, Virginia

REFERENCES:
- [Derived] Ehlers JP, Hu A, Boyer D, Cousins SW, Waheed NK, Rosenfeld PJ, Brown D, Kaiser PK, Abbruscato A, Gao G, Heier J; ReCLAIM-2 (SPIAM-202) Study Investigators. ReCLAIM-2: A Randomized Phase II Clinical Trial Evaluating Elamipretide in Age-related Macular Degeneration, Geographic Atrophy Growth, Visual Function, and Ellipsoid Zone Preservation. Ophthalmol Sci. 2024 Oct 9;5(1):100628. doi: 10.1016/j.xops.2024.100628. eCollection 2025 Jan-Feb. PMID 39605874

RESULTS

PARTICIPANT FLOW:
Groups:
- Elamipretide: 40 mg daily subcutaneous injection of elamipretide using the elamipretide delivery system for 48 weeks followed by a 4 week follow-up period.
- Placebo: Daily subcutaneous injection of placebo using the elamipretide delivery system for 48 weeks followed by a 4 week follow-up period.
Period: Overall Study
Arm/Group | Elamipretide | Placebo
Started | 117 | 59
Completed | 83 | 51
Not Completed | 34 | 8
Not completed — Withdrawal by Subject | 20 | 3
Not completed — Adverse Event | 10 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — COVID-19 infection | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were randomized and received at least one dose of study drug and have baseline and at least one post-baseline value for LL BCVA or GA Area on OCT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Elamipretide | Placebo | Total
Number analyzed (Participants) | 114 | 58 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (8.40) | 75.8 (8.80) | 76.0 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 36 | 104
  Male | 46 | 22 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 111 | 53 | 164
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 112 | 57 | 169
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 114 | 58 | 172
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: All individuals for whom body mass index was measured.
  kg/m^2
    number analyzed (Participants) | 111 | 57 | 168
    (all) | 29.85 (6.479) | 27.92 (5.380) | 29.20 (6.181)
GA Area (mm2) by OCT [Mean (Standard Deviation); unit: mm^2] | 1.47 (0.761) | 1.38 (0.682) | 1.44 (0.734)
LL BCVA Score [Mean (Standard Deviation); unit: Letters] — Low luminance best corrected visual acuity (LL BCVA) score assessment uses the Early Treatment Diabetic Retinopathy Study (ETDRS) scale. ETDRS charts present a series of letters of equal difficulty on each row with a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Scores range from 0-100. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
  Letters | 53.4 (16.17) | 58.8 (10.70) | 55.2 (14.75)
BCVA Score [Mean (Standard Deviation); unit: Letters] — Best corrected visual acuity (BCVA) score assessment uses the Early Treatment Diabetic Retinopathy Study (ETDRS) scale. ETDRS charts present a series of letters of equal difficulty on each row with a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Scores range from 0-100. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
  Letters | 75.8 (9.09) | 76.6 (7.90) | 76.1 (8.69)

OUTCOME MEASURES:

1. Primary Outcome: LL BCVA Score Change From Baseline
Description: Change in low luminance best corrected visual acuity (LL BCVA) score from Baseline to the end of treatment (EOT; Week 48) assessment measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale. ETDRS charts present a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows; there is a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Minimum score of zero, maximum score of 100. Change from baseline: a more negative score is worse outcome, a more positive score is better outcome. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
Time Frame: Baseline and Weeks 4, 8, 12, 24, 36, 48
Population: All subjects for which LL BCVA score change from Baseline was measured. All subjects were randomized and received at least one dose of study drug and have baseline and at least one post-baseline value for LL BCVA or GA Area on OCT. There was early study discontinuation for some of the participants and row numbers, including Week 4, reflect this.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 114 | 58
Letters
  Week 4: number analyzed (Participants) | 109 | 56
  Week 4 | 0.7 (6.11) | -0.6 (5.93)
  Week 8: number analyzed (Participants) | 103 | 54
  Week 8 | 1.1 (5.64) | -0.8 (7.71)
  Week 12: number analyzed (Participants) | 101 | 54
  Week 12 | -0.7 (9.35) | -0.9 (7.05)
  Week 24: number analyzed (Participants) | 93 | 52
  Week 24 | -0.9 (9.05) | -0.9 (6.80)
  Week 36: number analyzed (Participants) | 81 | 52
  Week 36 | -0.6 (12.21) | -3.2 (9.37)
  Week 48: number analyzed (Participants) | 82 | 48
  Week 48 | -2.8 (11.40) | -4.6 (11.89)

2. Primary Outcome: GA Area Change From Baseline by OCT
Description: Geographic atrophy (GA) area: change from baseline as measured by optical coherence tomography (OCT) from Baseline to the end of treatment (EOT; Week 48)
Time Frame: Baseline and Weeks 12, 24, 36, 48
Population: All subjects for which GA Area Change From Baseline by OCT was measured. All subjects were randomized and received at least one dose of study drug and have baseline and at least one post-baseline value for LL BCVA or GA Area on OCT. There was early study discontinuation for some of the participants and row numbers, including Week 12, reflect this.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 111 | 57
mm^2
  Week 12: number analyzed (Participants) | 98 | 50
  Week 12 | 0.082 (0.0889) | 0.071 (0.0812)
  Week 24: number analyzed (Participants) | 89 | 48
  Week 24 | 0.166 (0.1391) | 0.166 (0.1426)
  Week 36: number analyzed (Participants) | 75 | 47
  Week 36 | 0.245 (0.1680) | 0.228 (0.1977)
  Week 48: number analyzed (Participants) | 76 | 45
  Week 48 | 0.328 (0.2166) | 0.281 (0.2407)

3. Secondary Outcome: LL RA Change From Baseline
Description: Low-luminance ready acuity (LL RA) score change from baseline to the EOT (Week 48). Mean Critical Print Size with Low Luminance in Weeks 4, 12, 36, 48 as measured by the Logarithm of the Minimum Angle of Resolution LogMAR chart. Scores range from -0.3 to 1.0, where higher number means worse acuity/worse outcome, a lower number means better acuity/better outcome.
Time Frame: Baseline and Weeks 4,12, 36, 48
Population: All subjects for which LL RA change from baseline was measured. There was early study discontinuation for some of the participants and row numbers, including Week 4, reflect this.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 114 | 58
units on a scale
  Week 4: number analyzed (Participants) | 108 | 57
  Week 4 | -0.005 (0.2678) | 0.029 (0.3169)
  Week 12: number analyzed (Participants) | 100 | 53
  Week 12 | -0.008 (0.3429) | 0.035 (0.3244)
  Week 36: number analyzed (Participants) | 76 | 48
  Week 36 | 0.002 (0.3776) | 0.073 (0.2761)
  Week 48: number analyzed (Participants) | 82 | 48
  Week 48 | 0.011 (0.4082) | 0.101 (0.3069)

4. Secondary Outcome: BCVA Change From Baseline
Description: Best-corrected visual acuity (BCVA) change from Baseline Change in best corrected visual acuity (BCVA) score from Baseline to the end of treatment (EOT; Week 48) assessment measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale. ETDRS charts present a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows; there is a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Minimum score of zero, maximum score of 100. Change from baseline: a more negative score is worse outcome, a more positive score is better outcome. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
Time Frame: Baseline and Weeks 4, 8, 12, 24, 36, 48
Population: All subjects for which BCVA change from baseline was measured. There was early study discontinuation for some of the participants and row numbers, including Week 4, reflect this.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 114 | 58
Letters
  Week 4: number analyzed (Participants) | 109 | 57
  Week 4 | 0.3 (4.03) | -0.1 (4.51)
  Week 8: number analyzed (Participants) | 104 | 55
  Week 8 | 0.0 (4.88) | 0.9 (4.84)
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.2 (4.46) | -0.0 (6.14)
  Week 24: number analyzed (Participants) | 94 | 52
  Week 24 | -0.2 (5.09) | -0.2 (5.00)
  Week 36: number analyzed (Participants) | 81 | 52
  Week 36 | -1.5 (5.76) | -0.8 (6.13)
  Week 48: number analyzed (Participants) | 82 | 49
  Week 48 | -3.0 (6.90) | -2.6 (7.86)

5. Secondary Outcome: GA Area as Measured by Fundus Autofluorescence (FAF) Change From Baseline
Description: Change from Baseline in Mean Area of Geographic Atrophy (GA) by Fundus Autofluorescence (FAF) at Week 24. Fluorescein angiography (FA) was used to examine the circulation of the retina and choroid using fluorescein dye and a specialized camera to trace the dye. Fundus autofluorescence imaging of the retinal pigment epithelium and neurosensory retina was performed within 14 days of Day 0 and at every visit with the exception of Day 0 and Day 7. Atrophy is characterized by loss of the retinal pigment epithelium (RPE), overlying photoreceptors and underlying choriocapillaris. Greater area affected means a worse outcome than smaller area affected.
Time Frame: Baseline and Weeks 12, 24, 36, 48
Population: All subjects for which GA area as measured by fundus autofluorescence (FAF) change from baseline was measured. There was early study discontinuation for some of the participants and row numbers, including Week 12, reflect this.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 114 | 58
mm^2
  Week 12: number analyzed (Participants) | 98 | 50
  Week 12 | 0.074 (0.0690) | 0.065 (0.0804)
  Week 24: number analyzed (Participants) | 92 | 48
  Week 24 | 0.161 (0.1218) | 0.138 (0.1338)
  Week 36: number analyzed (Participants) | 77 | 50
  Week 36 | 0.242 (0.1659) | 0.199 (0.1700)
  Week 48: number analyzed (Participants) | 80 | 45
  Week 48 | 0.318 (0.2060) | 0.277 (0.2176)

6. Other Pre Specified Outcome: Macular Percentage of Ellipsoid Zone (EZ) Total Attenuation From Baseline
Description: Change from Baseline in Macular Percentage of EZ Total Attenuation by OCT: Week 24 and Week 48 measures photoreceptor loss marked by EZ degradation. Lower increase in percentage means a better outcome. Higher increase in percentage means a worse outcome.
Time Frame: Baseline, Week 24 and Week 48
Population: All subjects for which Macular Percentage of Ellipsoid Zone (EZ) Total Attenuation was measured. There was early study discontinuation for some of the participants and row numbers, including Week 24, reflect this.
Measure: Mean (Standard Deviation); unit: percentage of EZ total attentuation
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 114 | 58
percentage of EZ total attentuation
  Week 24: number analyzed (Participants) | 89 | 50
  Week 24 | 1.81 (3.889) | 2.70 (3.291)
  Week 48: number analyzed (Participants) | 71 | 42
  Week 48 | 3.94 (4.052) | 6.38 (6.616)

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Arm/Group | Elamipretide | Placebo
All-Cause Mortality (participants affected / at risk) | 2/117 | 0/59
Serious Adverse Events (participants affected / at risk) | 18/117 | 6/59
Other Adverse Events (participants affected / at risk) | 83/117 | 36/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elamipretide (N=117) | Placebo (N=59)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Corona virus infection (Infections and infestations) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elamipretide (N=117) | Placebo (N=59)
Injection Site Pruritus (General disorders) | 46 | 0
Injection Site Pain (General disorders) | 33 | 6
Injection Site Bruising (General disorders) | 15 | 11
Injection Site Erythema (General disorders) | 22 | 0
Injection Site Haemorrhage (General disorders) | 17 | 4
Injection Site Induration (General disorders) | 16 | 3
Injection Site Hypertrophy (General disorders) | 10 | 4
Injection Site Mass (General disorders) | 13 | 0
Injection Site Swelling (General disorders) | 11 | 0
Injection Site Irritation (General disorders) | 5 | 0
Injection Site Urticaria (General disorders) | 5 | 0
Injection Site Discomfort (General disorders) | 2 | 2
Neovascular Age-related Macular Degeneration (Eye disorders) | 8 | 5
Vitreous Floaters (Eye disorders) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 4 | 7
Pneumonia (Infections and infestations) | 4 | 1
Corona Virus Infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2
Headache (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Eosinophil Count Increased (Investigations) | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypertension (Vascular disorders) | 5 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03891875/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT03891875/SAP_001.pdf